CLINICAL TRIAL: NCT05302999
Title: Feasibility of Early Gabapentin as an Intervention for Neurorecovery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kimberly Anderson, PhD, Director, Northeast Ohio Regional SCI Model System, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB21-00609
Record Dates: First submitted 2022-02-22; First posted 2022-03-31 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries
Keywords: Gabapentin; Neurorecovery; Feasibility
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Low dose (Experimental): 600mg treatment group will receive 2 capsules of gabapentin by mouth 3 times per day for 90 days.
  Interventions: Drug: Gabapentin
- Medium dose (Experimental): 1800 mg treatment groups will receive 2 capsules of gabapentin by mouth 3 times per day for 90 days.
  Interventions: Drug: Gabapentin
- Control (Placebo Comparator): The control group will receive 2 placebo capsules of inert cellulose by mouth 3 times per day for 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Generic gabapentin
  Arms: Low dose; Medium dose
Drug: Placebo — Inert cellulose
  Arms: Control

SUMMARY:
The objective of the proposed study is to conduct the first ever prospective, dose-exploration trial to test the feasibility of early administration of gabapentin as an intervention for neurorecovery. This research project falls under the Intervention Development stage of research as the primary goal is to assess the feasibility of conducting a well-designed intervention efficacy study in the future.

DETAILED DESCRIPTION:
Gabapentin is a medication commonly used in spinal cord injury (SCI) to manage neuropathic pain. Emerging preclinical and clinical evidence suggests that early initiation of low to medium doses of gabapentin and continued delivery for a range of 2 weeks to 4 months has a persistent, positive effect on motor and autonomic neurologic recovery. The objective of the proposed study is to conduct the first ever prospective, dose-exploration trial to test the early administration of gabapentin as an intervention for neurorecovery. A mock efficacy design will be employed. Participants will be stratified based on ASIA Impairment Scale (AIS) grade A-B or C-D and randomized to 1 of 3 arms. Study medication will be initiated within 5 days post-injury and administered for 90 days. Participants will be followed for an additional 90 days after stopping treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic SCI;
2. All levels of SCI;
3. All severities of SCI, AIS A-D;
4. Age 18 years and older.
5. Agree to participate and start study drug within 120 hours' post-injury.
6. Adequate cognition and communication to provide informed consent

Exclusion Criteria:

1. Presence of moderate/severe traumatic brain injury (TBI) as defined by Glasgow Coma Score (GCS) < 13 at 120 hours' post-injury.
2. Documented use of gabapentinoids at the time of injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited | During the first 120 hours post-injury
  Feasibility question - Can the target population be recruited?
  Feasibility measure - Number screened/month; number enrolled/month; reasons for not enrolling
  Quantitative benchmark of success - Screen an average of 4/month; Enroll an average of 1/month
Adherence rate to drug treatment protocol | Across 90 day treatment window
  Feasibility question - Can the drug treatment protocol be delivered?
  Feasibility measure - Proportion of enrolled who receive the full drug treatment protocol (placebo arm; two gabapentin dose arms); number of dosing deviations/arm; reasons for dosing deviations
  Quantitative benchmark of success - 70% enrolled in placebo arm receive full dosing protocol; 70% enrolled in each gabapentin arm receive full dosing protocol
Number of occurrences of unblinding | Across 6 month study duration per participant
  Feasibility question - Can the assessors remain blinded?
  Feasibility measure - Number of occurrences of unblinding; reasons for unblinding
  Quantitative benchmark of success - 5% or fewer occurrences of unblinding
Retention rate | Across 6 month study duration per participant
  Feasibility question - Will participants complete the study?
  Feasibility measure - Retention rate; reasons for dropout; proportion of planned assessments completed
  Quantitative benchmark of success - 70% of participants stay enrolled until the end of the study and complete 3 of the 4 assessment visits

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kimberly Anderson, PhD, Principal Investigator — Metrohealth Medical Center-Case Western Reserve University School of Medicine
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson JR, Doty S, Petitt JC, El-Abtah M, Francis JJ, Sharpe MG, Kelly ML, Anderson KD. Feasibility of gabapentin as an intervention for neurorecovery after an acute spinal cord injury: Protocol. Front Neurol. 2022 Nov 7;13:1033386. doi: 10.3389/fneur.2022.1033386. eCollection 2022. PMID 36419530